CLINICAL TRIAL: NCT06668246
Title: Performance of Refractometers With Self-adjusting Lenses Compared to Cycloplegia in Children
Brief Title: Performance of Refractometers With Self-adjusting Lenses Compared to Cycloplegia in Children (REFRALENS)
Acronym: REFRALENS
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0231 - REFRALENS
Record Dates: First submitted 2024-10-28; First posted 2024-10-31 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-09

CONDITIONS: Refractive Errors; Ametropia
MeSH Terms: conditions — Refractive Errors | interventions — Immersion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Vision-S™ 700, an immersive and compact phoropter with a tunable-focus lens, and Vision-R™ 800, a phoropter with a tunable-focus lens without immersion, with cycloplegic refraction serving as the gold — As of today, no published clinical studies have been conducted with the Vision-S™ 700 neither Vision R 800

SUMMARY:
This study aimed to compare refractive measurements using Vision-S™ 700, an immersive and compact phoropter with a tunable-focus lens, and Vision-R™ 800, a phoropter with a tunable-focus lens without immersion, with cycloplegic refraction serving as the gold-standard.

This a retrospective study aimed to enroll 41 children, aged 6 to 16 years, who underwent refractive assessments with Vision-S™ 700, Vision-R™ 800, and cycloplegic refraction. The primary objective involves a comparison of the spherical equivalent between both devices and compared to cycloplegic refraction. Secondary outcomes include the analysis of astigmatism components (J0° and J45°) and subgroup analyses in myopic and hyperopic children.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 16 years old patients followed in the Brest University Hospital Center, in France, between the 1st of November 2022 and the 30th of April 2023 and requiring a cycloplegic refraction not presenting an exclusion criteria

Exclusion Criteria:

* age below 6 years or above 16 years
* presence of other ophthalmological pathologies rather than ametropia
* non-French language proficiency, and absence of parental authorization

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 6 to 16 years old patients followed in the Brest University Hospital Center, in France, between the 1st of November 2022 and the 30th of April 2023 and requiring a cycloplegic refraction not presenting an exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 41 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Spherical equivalent | Day 1
  The primary outcome of this study was to compare the spherical equivalent, obtained using two different devices: Vision-S™ 700, an immersive phoropter with a tunable-focus lens, and Vision-R™ 800, a phoropter with a tunable-focus lens without immersion. The study aimed to assess the overall agreement of these measurements with cycloplegic refraction, considered the gold standard in this context.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement